CLINICAL TRIAL: NCT01833013
Title: Infertility and Endometriosis : a Prospective Cohort Study
Brief Title: Infertility and Endometriosis Cohort
Acronym: EndoFertil
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 9113
Record Dates: First submitted 2013-04-11; First posted 2013-04-16 (Estimated); Last update posted 2015-01-09 (Estimated); Status verified 2013-04

CONDITIONS: Endometriosis; Infertility
Keywords: Endometriosis; Cohort study; fertility; pregnancy; assisted reproductive technics; laparoscopy
MeSH Terms: conditions — Endometriosis; Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- endometriosis cohort (Other): females suffer from endometriosis
  Interventions: Other: live birth date and quality of life assessment

INTERVENTIONS:
Other: live birth date and quality of life assessment

SUMMARY:
Nowadays, one in six couples consults for fertility problems. If the standard examination and tests do not reveal any cause of infertility, the woman may undergo a laparoscopic exploration which reveals endometriosis in more than 50% of cases.

Endometriosis is an inflammatory disease defined as the presence of endometrial tissue out of the uterine cavity. It is frequent (1 in 10 women) and associated with a high economic burden (22 billion dollars in 2002 in the USA) and important decrease in quality of life. Physiopathological mechanisms and risk factors for endometriosis are not well identified.

A woman with endometriosis is 20 times more at risk of infertility. Fecundity rate of a 25-year-old couple is about 15 to 20% in the general population and only 2 to 10% in case of endometriosis.

There are many manifestations of this disease (infertility, pelvic pain) and the anatomo-clinical correlation is not good. The presently used international classification (American Fertility Society revised in 1985, AFSr) does not predict the chance of pregnancy. New scores such as the Endometriosis Fertility Index (EFI) have been proposed to do so, but need to be validated. Treatment for endometriosis-related infertility is not consensual.

A prospective cohort study would give access to clinical data of patients followed in our center, so as to identify clinical factors predicting pregnancy and to help treatment decision for women with endometriosis suffering from infertility.

ELIGIBILITY:
Inclusion criteria:

* Woman from 18 to 41 years old.
* Dealing with infertility,
* With a normal pelvic echography and hysterosalpingography, a normal hormonal status and a partner with a normal sperm.
* For whom a laparoscopic exploration finds endometriosis.
* Consenting to participate to the study.

Exclusion criteria:

* Any contraindication for general anesthesia or for laparoscopy.
* Any contraindication for pregnancy.
* Follow-up is impossible.
* Consent is impossible.

Ages: 18 Years to 41 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2013-04; Primary Completion 2018-04 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
live birth date | 3 years
  Assessment of the number of live birth in the 3 years following the laparoscopic exploration making the diagnosis of endometriosis

SECONDARY OUTCOMES:
Quality of life | 3 years
  Assessment of the quality of life relating to infertility and endometriosis in the 3 years following laparoscopic exploration making the diagnosis of endometriosis.
pain symptoms | 3 years
  Assessment of the pain symptoms relating to infertility and endometriosis in the 3 years following laparoscopic exploration making the diagnosis of endometriosis.

CONTACTS AND LOCATIONS:
Overall Officials: Herve Dechaud, MD,PhD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- University Hospital Montpellier, Montpellier, Herault, France